CLINICAL TRIAL: NCT01670682
Title: A Prospective，Multicenter Pilot Study to Compare Ischia Spinous Fascia Fixation Procedure With Modified Total Pelvic Floor Reconstruction Surgery For Pelvic Organ Prolapse Stage III
Brief Title: Ischia Spinous Fascia Fixation Procedure Versus Modified Total Pelvic Floor Reconstructive Surgery for Pelvic Organ Prolapse Stage III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pumch-gyn-03
Record Dates: First submitted 2012-02-22; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: Stage III
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fascia fixation group (Active Comparator): procedure: ischia spinous fascia fixation
  Interventions: Procedure: ischia spinous fascia fixation
- mesh group (Active Comparator): Procedure: Modified Pelvic Floor Reconstruction Surgery with mesh
  Interventions: Procedure: Modified Pelvic Floor Reconstruction Surgery with Mesh; Device: polypropylene mesh(Gynemesh)

INTERVENTIONS:
Procedure: ischia spinous fascia fixation — Subjects of this group were submitted to surgical treatment with ischia spinous fascia fixation.
  Arms: fascia fixation group
Procedure: Modified Pelvic Floor Reconstruction Surgery with Mesh — Subjects of this group were submitted to surgical treatment with Modified Total Pelvic Floor Reconstruction Surgery with Mesh.
  Arms: mesh group
Device: polypropylene mesh(Gynemesh) — Pelvic floor reconstruction will be conducted using surgical mesh made from polypropylene.
  Arms: mesh group

SUMMARY:
Pelvic organ prolapse is a common problem. The primary treatment is surgery. Ischia spinous fascia fixation procedure and modified total pelvic floor reconstructive surgery with mesh are both developed in China for vaginal apex fixation, the former is native tissue repairs, and the latter is augmentation with mesh.

This study is designed to determine the effectiveness and safety of ischia spinous fascia fixation procedure compared with modified total pelvic floor reconstructive surgery with mesh for the treatment of pelvic organ prolapse stage III.

Patients enrolled into the study will be followed up for up to 3 years after surgery. Evaluation will take place during surgery and postoperative visit. Stage of prolapse before and after surgery, patient satisfaction through quality of life and sexual function questionnaires before and after surgery, and peri-operative complication rates will be evaluated.

DETAILED DESCRIPTION:
Pelvic Organ prolapse (a feeling of bulge in the vagina) may cause some distressing symptoms such as loss of control of the bowel or bladder, and may also cause problems with patient's sex life. An ideal procedure for vaginal apical support should provide a durable suspension, have minimal complications, and not affect sexual or visceral function.

Vaginal procedures used for restoring the vaginal apex support include Ischia spinous fascia fixation procedure with native tissue and modified total pelvic floor reconstructive surgery with mesh. They are both developed and popular in China. Clinical practice showed that they were both safe, efficient and cost-effective. Recurrent rates of both procedures after 1 year follow-up were about 10%, and quality of life improved significantly from the baseline, while the.complications are different.

The purpose of this multicenter, prospective, and comparative study is to evaluate the effectiveness and safety of these two procedures in the treatment of symptomatic pelvic organ prolapse Stage III in China.

ELIGIBILITY:
Inclusion Criteria:

* Candidates with symptomatic pelvic organ prolapse of POP-Q Stage III, suitable for surgical repair.
* Vaginal hysterectomy and anti-incontinence procedures could be performed concurrently.
* Age ≥ 55 years.
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires.

Exclusion Criteria:

* Previous repair of pelvic organ prolapse involving insertion of mesh.
* Experimental drug or experimental medical device within 3 months prior to the planned procedure.
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Coagulation disorder or on therapeutic anticoagulant therapy at the time of surgery.
* History of chemotherapy or pelvic radiation therapy.
* Systemic disease known to affect bladder or bowel function (e.g. Parkinson's disease, multiple sclerosis, spinal cord injury or trauma).
* Current evaluation or treatment for chronic pelvic pain (e.g. interstitial cystitis, endometriosis, coccydynia, vulvodynia).
* Nursing or pregnant or intends future pregnancy.
* Chronic cough not well-controlled.
* BMI ≥ 30.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
•Anatomical improvement according to POP-Q score. | 6 weeks
•Anatomical improvement according to POP-Q score. | 1 year
•Anatomical improvement according to POP-Q score. | 2 years
•Anatomical improvement according to POP-Q score. | 3 years

SECONDARY OUTCOMES:
•Hospital data including operative time, estimated blood loss, length of stay, maximum temperature, time of voiding recovery. | At discharge, an expected average of 5 days after operation.
•Pain score measured using Visual Analog Scale (VAS). | 24 hours post surgery and at the 6-week visit
•Presence/absence of complications (composite score). | Up to 6 weeks.
  The occurrence (in the per-operative phase or within 6 weeks post-op) of at least one of the following: 1) bleeding complications; 2) infectious complications; 3) any wound caused by a surgeon movement: bladder, ureteral, or vascular injuries; 4)medical complications: deep vein thrombosis, pulmonary embolism and etc.Complications will be categorized using the Dindo surgical complication grading scale.
•Change from baseline in PFIQ-7 scores. | 1 year, 2 years and 3 years.
•In subjects sexually active at baseline, assessment of sexual function using PISQ-12 (mean scores and change from baseline) | 1 year, 2 years and 3 years.
•Subject global impression assessed on a 5 point Likert scale | 1 year, 2 years and 3 years.
•Presence/absence of complications (composite score) | Up to 3 years.
  Long-term negative outcomes of the surgical procedure will also be recorded until 3 years after surgery. For example, mesh erosion, de novo urinary incontinence, de novo dyspareunia and overall failure rate. Complications will be categorized using the Dindo surgical complication grading scale.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Foshan Maternal and Child Health Hospital, Foshan, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - the Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Affiliated Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Peking Union Medical College Hospital, Beijing